CLINICAL TRIAL: NCT00887263
Title: Double-blind, Randomised, Placebo-controlled Multicentre Phase III Clinical Study Followed by Open-label Phase on the Efficacy and Tolerability of Budesonide 3 mg Effervescent Tablet in Patients With Resistant Oral Chronic GvHD
Brief Title: Efficacy and Safety Study of Budesonide to Treat Oral Chronic Graft vs Host Disease (cGvHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUM-5/GVH
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Oral Chronic Graft vs Host Disease
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Budesonide
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — 3 mg TID
  Arms: A
Drug: Placebo — 0 mg TID
  Arms: B

SUMMARY:
The purpose of the study is to compare the efficacy and tolerability of budesonide 3 mg effervescent tablet (9 mg/day) compared to placebo for the treatment of patients with resistant oral cGvHD.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky >= 70
* Oral chronic GvHD after allogeneic haematopoietic stem cell transplantation
* Oral cGvHD of erosive and/or ulcerative type
* NIH scale >= 3
* Resistant oral cGvHD with no oral response to conventional primary treatment

Exclusion Criteria:

* Uncertain diagnosis of resistant oral cGvHD
* Symptomatic oral cGvHD of hyperkeratotic type solely
* Current active oral bacterial, viral, or fungal infection
* Unwilling to forego concurrent treatment for mucosal lesions and/or related oral pain
* Requiring addition of new systemic therapy including steroids, or radiation therapy
* Local intestinal infection
* Abnormal hepatic function or liver cirrhosis
* If careful medical monitoring is not ensured: tuberculosis, cardiovascular disease, diabetes mellitus, osteoporosis, active peptic ulcer disease, glaucoma, cataract, infection
* Second line treatment of oral cGvHD with topical steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2009-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of patients with objective response | 12 weeks

SECONDARY OUTCOMES:
Rate of complete/partial response, stable disease, progressive disease | 12 weeks
Time to initial objective response | x weeks
Rate of subjective improvement | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Elad, DMD, Principal Investigator — University of Rochester Medical Center, Division of Oral Medicine, Eastman Institute for Oral Health
Locations (2):
- University of Regensburg, Regensburg, Germany
- The Hebrew University-Hadassah School of Dental Medicine, Department of Oral Medicine, Jerusalem, Israel

REFERENCES:
- [Background] Elad S, Or R, Garfunkel AA, Shapira MY. Budesonide: a novel treatment for oral chronic graft versus host disease. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Mar;95(3):308-11. doi: 10.1067/moe.2003.23. PMID 12627101
- [Derived] Elad S, Zeevi I, Finke J, Koldehoff M, Schwerdtfeger R, Wolff D, Mohrbacher R, Levitt M, Greinwald R, Shapira MY. Improvement in oral chronic graft-versus-host disease with the administration of effervescent tablets of topical budesonide-an open, randomized, multicenter study. Biol Blood Marrow Transplant. 2012 Jan;18(1):134-40. doi: 10.1016/j.bbmt.2011.06.001. Epub 2011 Jun 12. PMID 21703973